CLINICAL TRIAL: NCT02904213
Title: A Bridging Study to Evaluate Safety of ComBe Five (Liquid) (Combined Pentavalent DTwP-rHepB-Hib Vaccine) Made in India, in Healthy Vietnamese Children Aged From 8 - 10 Weeks as a 3-dose Series, Interval for Each Dose is 4 Weeks
Brief Title: Evaluate Safety of ComBe Five (Liquid) in Healthy Vietnamese Children Aged From 8 - 10 Weeks as a 3-dose Series, Interval for Each Dose is 4 Weeks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Clinical Research and Clinical Trial Support for Vaccine and Biological Products (Other)
Collaborators: Biological E. Limited (Unknown)
Responsible Party: Principal Investigator, Pham Ngoc Hung, Principal Investigator, Vietnam Military Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VX.2016.03
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Safety, Pentavalent Vaccine
Keywords: vaccine; ComBe Five; Vietnam; pentavalent
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pentavalent vaccine (Experimental): 3 Dose, interval for each dose is 4 weeks. The first dose will be received at 8-10 weeks of age
  Interventions: Biological: ComBe Five (Liquid)

INTERVENTIONS:
Biological: ComBe Five (Liquid)

SUMMARY:
An open label, non-comparative bridging study to evaluate the safety of pentavalent vaccine ComBe Five (Liquid) made in India, in healthy Vietnamese children aged from 8 - 10 weeks as a 3-dose series, interval for each dose is 4 weeks

DETAILED DESCRIPTION:
The trial is a bridging Study to evaluate safety of pentavalent vaccine ComBe Five (Liquid) made in India, in healthy Vietnamese children aged from 8 - 10 weeks as a 3-dose series, interval for each dose is 4 weeks. 330 subjects will be enrolled in Binh Luc and Ly Nhan district, Ha Nam province. These subjects will be received 3 doses (0.5ml/dose) ComBe Five (Liquid), the first dose will be administered at 8-10 weeks of age.

The frequency, rate and severity of immediate adverse events within 30 minutes after vaccination, solicited and unsolicited AE within 28 days after vaccination, the frequency and rate of SAE within 28 days after the first vaccination will be recorded as evidences for ComBeFive (Liquid) safety assessment. The subjects to be included from this trial would be representative of the population of Vietnam.

The protocol has been reviewed and approved by Vietnam Military Medical University IRB and Vietnam Ministry of Health IEC and Vietnam Minister of Health.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all criteria below to participate in study:

1. Healthy children, both genders, age from 8 -12 weeks at screening visit and the first dose (visit 1)
2. Weight ≥ 3.300 gram at Screening visit and receive the first dose
3. Understand and follow the study
4. Mother of children have serum negative for HIV, HBV and HCV on blood test results or antenatal tests report book.
5. Children or mother don't participate in other clinical study scheduled during the study.
6. Parent/ legal guardian can understand and have ability to follow protocol.
7. Parent/ legal guardian voluntary write consent to participate in the study.
8. Parent/ legal guardian of subject have ability to comply with the process of study.
9. Parent/ legal guardian of subject who intends to remain in the area with the participant during the study period.

Exclusion Criteria:

Subject have one of criteria below must not participate in study:

1. Fever (temperature ≥37.5oC) or loses temperature (≤35.5 oC) or disease/ infection chronic
2. Subjects who had received DPT
3. Subjects who had received immunosuppressant therapy
4. Subjects with a known or doubt hypersensitivity of allergic reaction to any component of the study vaccine
5. Subjects who had any signs or symptoms of functional disorder, especially central nervous system.
6. Subjects who had haemophilia or received treatment anticoagulant drug, had a risk of serious bleeding when intramuscular injection.
7. Subjects who had a family history of SIDS (Sudden Infant death syndrome)
8. Subjects intend to surgery scheduled during the study
9. Subjects who had received any blood products, corticosteroid cytotoxic drugs, radiotherapy.
10. Subjects and mother who had participated in other clinical trial within 30 days priors to vaccination with study drug, or those who had another clinical trial scheduled during the study.
11. Can't afford or not ready follow protocol
12. Any criteria that, in the judgment of the investigator, would interfere with or serves as a contraindication to protocol adherence

Ages: 8 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2016-12-19 (Actual); Study Completion 2017-06-24 (Actual)

PRIMARY OUTCOMES:
Frequency and rate of the adverse effects and severity of immediate adverse events (Local and General) within 30 minutes after vaccination. | 30 minutes after vaccination
Frequency and rate of adverse effects and severity of solicited adverse events (Local and General) within 7 days after each vaccination | For 7 days after each vaccination
Frequency and rate of adverse effects and severity of unsolicited adverse events (Local and General) during 28 days after each vaccination | For 28 days after each vaccination
Frequency and rate of adverse effects and severity of Serious Adverse Events (Local and General) during 28 days after each vaccination | For 28 days after each vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Ha Nam Health Center, Hà Nam, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided